CLINICAL TRIAL: NCT04358952
Title: Imaging Cardiac Phenotype of SARS-Cov-2 (Covid19) Infected Patients
Brief Title: Myocardial Involvement of Severe Acute Respiratory Syndrome-Cov-2 (Covid19) Infected Patients
Acronym: COCARDE
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0117; 2020-A00852-37 (Other: ID RCB)
Record Dates: First submitted 2020-04-09; First posted 2020-04-24 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Cardiomyopathies
Keywords: Left ventricular systolic function; left ventricular diastolic function; global longitudinal strain; SARS-Cov-2; Covid-19
MeSH Terms: conditions — Cardiomyopathies; COVID-19 | interventions — Global Longitudinal Strain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Inflammatory cytokines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID + patients: Major patients hospitalized for respiratory criteria for SARS-Cov-2 infection confirmed by RT-PCR
  Interventions: Diagnostic Test: Global Longitudinal Strain

INTERVENTIONS:
Diagnostic Test: Global Longitudinal Strain — Electrocardiogram with measure of the Global Longitudinal Strain to evaluate myocardiac dysfunction

SUMMARY:
The effects of severe acute respiratory syndrome SARS-Cov-2 (Covid-19) on the myocardium and their role in the clinical course of infected patients are still unknown. Epidemiological studies report biological myocardial involvement in 10 to 25% of cases. The objective of this study is to cardiac phenotype using comprehensive cardiac imaging tools of patients infected with Covid 19 in order to explore the functional impact of the infection on the myocardium.

DETAILED DESCRIPTION:
A large population of Covid 19 infected patients of different ages and severity levels will be explored by transthoracic echocardiography with measurement of myocardial functional parameters such as ejection fraction, longitudinal strain and relaxation parameters and will be compared to an uninfected population paired for age and sex.

Patients with biological myocardial involvement will be followed to determine the evolution of their myocardial functional parameters during the course of the infection.

ELIGIBILITY:
Inclusion Criteria:

* Major patients hospitalized for respiratory criteria for SARS-Cov-2 infection confirmed by RT-PCR

Exclusion Criteria:

* Underage patients. Patients refusing to participate in research. Patients with a history of heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients hospitalized for respiratory criteria for SARS-Cov-2 infection confirmed by RT-PCR
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Left ventricular function | Day 0
  Left ventricular function evaluated by global longitudinal strain
Left ventricular function | Day 3
  Left ventricular function evaluated by global longitudinal strain
Left ventricular function | Day 7
  Left ventricular function evaluated by global longitudinal strain

SECONDARY OUTCOMES:
inflammatory biological parameters | Day 0
  Cytokine rate

CONTACTS AND LOCATIONS:
Overall Officials: Vincent MINVILLE, PU-PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

REFERENCES:
- [Derived] Lairez O, Blanchard V, Balardy L, Vardon-Bounes F, Cazalbou S, Ruiz S, Collot S, Houard V, Rolland Y, Conil JM, Minville V. COCARDE Study-Cardiac Imaging Phenotype in Patients With COVID-19: Protocol for a Prospective Observational Study. JMIR Res Protoc. 2022 Jan 6;11(1):e24931. doi: 10.2196/24931. PMID 34751159